CLINICAL TRIAL: NCT06568809
Title: Timing of Surgery in Pediatric Patients Following Fever Recovery: a Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Lu Yi, physician-in-charge, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2024-03-216
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-03

CONDITIONS: Fever
Keywords: Fever; SARS-CoV-2; Hypoxemia; Children
MeSH Terms: conditions — Fever; Hypoxia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 0-2 weeks; 3-4 weeks; 5-6 weeks; 7-8 weeks: The time between body temperature recovery and surgery was collected as categorical factor and was scheduled to be analyzed in the following categories: 0-2 weeks; 3-4 weeks; 5-6 weeks; 7-8 weeks.
  1. Before operation:
     ① Ask the children about the history of upper respiratory tract infection complicated with fever, and record the symptoms of upper respiratory tract infection.
     ② The symptoms of upper respiratory tract infection were collected on the day of operation.
     ③ Record the patient's age, sex, height, weight and ASA grade.
     ④ The preoperative chest X-ray imaging examination was collected.
  2. During the operation:
     * Record the average arterial pressure and heart rate before and after entering the room, intubation, extubation and operation room.
       ② Record the lowest value of oxygen saturation of hypoxemia during intubation and extubation.
       ③ Record the treatment process when PRAEs appear.
       ④ Record all anesthetic dosage.
       ⑤ Record the total operation time.
  Interventions: Other: Time interval between recovery of body temperature and operation
- ≥3 month(control group): The time between body temperature recovery and surgery was collected as categorical factor and was scheduled to be analyzed in the following categories≥ 3 months (control group).
  1. Before operation:
     ① Ask the children about the history of upper respiratory tract infection complicated with fever, and record the symptoms of upper respiratory tract infection.
     ② The symptoms of upper respiratory tract infection were collected on the day of operation.
     ③ Record the patient's age, sex, height, weight and ASA grade.
     ④ The preoperative chest X-ray imaging examination was collected.
  2. During the operation:
     * Record the average arterial pressure and heart rate before and after entering the room, intubation, extubation and operation room.
       ② Record the lowest value of oxygen saturation of hypoxemia during intubation and extubation.
       ③ Record the treatment process when PRAEs appear.
       ④ Record all anesthetic dosage.
       ⑤ Record the total operation time.
  Interventions: Other: Time interval between recovery of body temperature and operation

INTERVENTIONS:
Other: Time interval between recovery of body temperature and operation — The time between body temperature recovery and surgery was collected as categorical factor and was scheduled to be analyzed in the following categories: 0-2 weeks; 3-4 weeks; 5-6 weeks; 7-8 weeks; And ≥ 3 months (control group).

SUMMARY:
Objectives: The timing of fever recovery may affect the risk of intra-operative hypoxemia in children undergoing elective surgery after SARS-CoV-2 infection. This study aims to determine the optimal timing for surgery by analyzing the occurrence of intra-operative hypoxemia in pediatric patients after they have recovered from a fever.

Methods: This prospective cohort study included 3053 children who had been infected with SARS-CoV-2 and developed fever, and scheduled to a surgery during March 2023 to August 2023, children with temperature recovery time ≥3 month were compared to children with temperature recovery time 0-8weeks. The primary outcome was measured as the incidence of intra-operative hypoxemia in SARS-CoV-2 infected children after their body temperature returned to normal. Logistic regression models were used to calculate the adjusted incidence of hypoxemia rate sratified by time (0-2 weeks; 3-4 weeks; 5-6 weeks; 7-8 weeks; ≥3 month) from body temperature recovery to the day of surgery.

DETAILED DESCRIPTION:
This prospective cohort study included 3053 pediatric patients who had been infected with SARS-CoV-2 and developed fever, and scheduled to a surgery during March 2023 to August 2023.On the day of operation, the anesthesiologist in the children's operating room conducted a preoperative evaluation. Upon confirming that general anesthesia was appropriate, they proceeded to sign the informed consent for anesthesia. Three anesthesiologists were assigned to the research group and conducted a second preoperative visit to the children and their guardians in a separate room.

Body temperatures over 37.5 degrees Celsius was considered as fever. The time between body temperature recovery and surgery was collected as categorical factor and was scheduled to be analyzed in the following categories: 0-2 weeks; 3-4 weeks; 5-6 weeks; 7-8 weeks; And ≥ 3 months (control group). After entering the operating room, the children were routinely monitored (pulse oxygen saturation-SpO2, blood pressure and electrocardiogram). The anesthesia method and drug selection were decided by the anesthesiologist in the operating room. The following data were collected and recorded: age, height, weight and ASA classification; The preoperative medication and the perioperative use of narcotic drugs ; The induction technique; The primary airway device; The lowest value of SpO2 when the child entered the operating room, was intubated and was extubated; PRAEs (such as cough, wheezing, laryngeal spasm and bronchial spasm) occurred during operation; The treatment processwhen PRAEs occured; The total duration of operation. The primary outcome was the incidence of intra-operative hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

1) Pediatric patients aged 1 to 18 years old; 2) American Society of Anesthesiologists physical status (ASA) Ⅰ or Ⅱ; 3) Undergoing selective tonsillectomy, nasal and paranasal sinus surgery, inguinal hernia repair, circumcision, internal fixation removal and other elective or daytime operations in otolaryngology, general surgery or orthopedics.

Exclusion Criteria:

1) the weight is either less than or more than 15% of standard weight [standard weight (kg) = height (cm) -100]; 2) body mass index (BMI) < 13.5 kg/m2 or > 31 kg/m2; 3) presence of asthma or airway hyperresponsiveness, neuromuscular systemic disease or cachexia, or difficult airway; 4) abnormal surgical anesthesia recovery history; 5) operation duration > 2 hours; 6) participants in any drug clinical trial within 30 days before the study; 7) absence of a definite date of fever recovery and other conditions deemed unsuitable for inclusion by the researchers.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This prospective cohort study included 3053 pediatric patients who had been infected with SARS-CoV-2 and developed fever, and scheduled to a surgery during March 2023 to August 2023. Body temperatures over 37.5 degrees Celsius was considered as fever. The patient's guardian provided the recovery date of the child's fever. The time between body temperature recovery and surgery was collected as categorical factor and was scheduled to be analyzed in the following categories: 0-2 weeks; 3-4 weeks; 5-6 weeks; 7-8 weeks; And ≥ 3 months (control group).
Sampling Method: Non-Probability Sample
Enrollment: 3053 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Pulse oxygen saturation | intubation, extubation and operation
  Record the lowest oxygen saturation of hypoxemia during intubation, extubation and operation.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yi, physician, Principal Investigator — The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided